CLINICAL TRIAL: NCT05877664
Title: A Phase 1 Dose Escalation and Expansion, Tolerability, Safety, Pharmacokinetics / Pharmacodynamics and Preliminary Efficacy Study of ZG0895.HCl in Patients With Advanced Solid Tumors
Brief Title: Study of ZG0895.HCl in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZG0895-001
Record Dates: First submitted 2023-05-11; First posted 2023-05-26 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Part1：Dose Escalation (Experimental): During the dose-escalation stage, an accelerated titration design (ATD) will be utilized for the first three lower dose groups (0.06, 0.12 and 0.18 mg/m^2). The conventional "3+3" dose escalation method will be used for the subsequent dose groups. The entire duration of 21 days after the first dose of ZG0895.HCl is defined as the dose-limiting toxicity (DLT) observation period.
  Interventions: Drug: ZG0895 Hydrochloride for Injection

INTERVENTIONS:
Drug: ZG0895 Hydrochloride for Injection — The dose escalation of ZG0895.HCl is set as 0.06, 0.12, 0.18, 0.37, 0.75, 1.50, 2.25, 3.00, and 3.75 mg/m^2 groups, subcutaneous (SC) injection once a week (QW)
  Other Names: ZG0895.HCl

SUMMARY:
The primary objective of this study is to assess the tolerability and safety of ZG0895.HCl, and to assess the maximum tolerated dose (MTD)/ recommended phase 2 dose (RP2D) of ZG0895.HCl.

ELIGIBILITY:
Inclusion Criteria:

* Fully understand the study and voluntarily sign the informed consent form(ICF).
* Age ≥ 18 and ≤ 75 years old at the time of signing the ICF, either male or female;
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
* Life expectancy ≥ 3 months.
* All adverse events from prior treatment have either returned to baseline or CTCAE 5.0 ≤ Grade 1(except for AEs not constituting a safety risk in the opinions of the investigators, e.g. alopecia, hypothyroidism which can be treated with a hormone replacement, etc).
* Both male and female participants (unless postmenopausal, surgical sterilization) and partners must agree to use a reliable form of contraception during the study treatment period and for at least 6 months after the last dose of the study drug.
* For lesions that have received radiation therapy, only after the progression of the lesions, they can be considered measurable lesions.

Part 1:

* Must have at least 1 measurable lesion per Response Evaluation Criteria in Solid Tumors v1.1 (RECIST v1.1).
* Participants with histologically or cytologically confirmed diagnosis of advanced solid tumors, in whom available standard treatments failed or were intolerable.

Exclusion Criteria:

* Participants receiving any of the following treatments:

  1. Previously treated with systemic TLR7/8 immunomodulators.
  2. Any other investigational product treatment within 4 weeks before the first dosing.
  3. Chemotherapy, biotherapy, endocrine therapy (except for hormone replacement), and biological targeted medicines within 4 weeks before the first dosing. Local palliative radiotherapy, traditional Chinese medicine with anti-tumor effect, and small molecule targeted therapy within 2 weeks (or 5 half-lives, whichever is longer) before the first dosing.
  4. Major surgery within 4 weeks before the first dosing for any reason (excluding puncture biopsy), or need to undergo elective surgery during the trial.
  5. Potent CYP3A4/5 inducer or inhibitor within 2 weeks prior to administration of the first dose of the study drug.
  6. Systemic immunosuppressive drugs within 2 weeks prior to administration of the first dose of the study drug, including systemic corticosteroids (>10 mg/day prednisone or equivalent).
  7. Other immunomodulators within 2 weeks prior to administration of the first dose of the study drug, including but not limited to thymosin, interleukin-2 and interferon.
* Had CTCAE Grade ≥3 immune-related adverse events (irAE) after receiving immunotherapy.
* The main organ function meets any of the following criteria within 7 days prior to the first dosing. （Note: blood transfusion, EPO, G-CSF, albumin infusion and renal replacement therapy are not allowed within 14 days prior to treatment.)

  1. Hematological function: ANC < 1.5×10^9/L, PLT < 75×10^9/L, Hemoglobin (Hb) < 100 g/L.
  2. Hepatic function: Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≥ 3×ULN; ALT and AST ≥ 5×ULN for participants with liver metastases; Total bilirubin (TBIL) ≥ 1.5×ULN; albumin < 30 g/L.
  3. Creatinine clearance< 75 mL/min.
  4. INR > 1.5 or APTT > 1.5×ULN.
  5. The urine protein presents positive and the quantitative result of 24-h urine protein ≥ 1 g.
* Participants with symptomatic central nervous system (CNS) metastases or carcinomatous meningitis; or other evidence suggesting that the central nervous system metastasis or meningeal metastasis is not well-controlled and is judged by the investigator to be unsuitable for enrollment.
* Uncontrollable third cavity effusion (e.g. large amount pleural effusion, ascites, or pericardial effusion, etc.) requiring repeated drainage, which is judged by the investigator to be unsuitable for enrollment.
* Known history of neurological disorders affecting brain functional activities, including epilepsy or dementia.
* Severe cardiac-cerebral vascular disease, including but not limited to:

  1. Acute myocardial infarction, unstable angina, stroke, or received coronary angioplasty or stent implantation within 6 months before the first dosing.
  2. New York Heart Association functional class II to IV congestive heart failure or left ventricular ejection fraction (LVEF) < 50% or the lower normal limit.
  3. Uncontrollable hypertension (even though the best available treatment is used but systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg).
  4. QTcF interval prolongation during the baseline period.
* Participants with active or history of autoimmune diseases (such as systemic lupus erythematosus, rheumatoid arthritis, vasculitis, etc.), except for clinically stable autoimmune thyroid diseases.
* Active infection requiring systemic therapy within 7 days prior to the first dosing; active hepatitis B or hepatitis C, history of immunodeficiency virus (HIV) disease or HIV antibody positive.
* Priorly received allogeneic stem cell transplantation or solid organ transplantation.
* Known allergy to the ZG0895.HCl or any of its excipients; have severe allergy history (CTCAE Grade ≥ 3), such as severe urticaria, angioedema, severe anaphylaxis, etc.
* Females who are pregnant or nursing during the screening period.
* The investigators consider that the participants are not suitable to participate in the clinical study for other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08-08 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
The incidence of dose-limiting toxicity (DLT) | Up to Day 21
  DLT is defined as any of the following adverse events (AE) occurring from the first dose of Day 1 to Day 21, unless the investigator deems that the AE is clearly related to the disease progress or definitely due to an external cause. Delayed DLTs are adverse events that meet the criteria of DLTs that occur after Cycle 1. All AEs will be graded according to the US National Cancer Institute Common Terminology Criteria for Adverse Events Version 5.0 (NCI CTCAE v5.0), except for cytokine release syndrome (CRS)
The maximum tolerated dose (MTD) of ZG0895.HCl | Up to Day 21
  During the dose-escalation stage, if there is a first occurrence that ≥ 2 participants in a dose group experience DLT, then the dose level will be considered to be an intolerable dose, and the previous lower dose will be considered to be the MTD. The MTD group should have at least 6 evaluable participants.
Number of Participants Experiencing Adverse Events (AEs) | Up to 3 Years
Number of Participants Experiencing Serious Adverse Events (SAEs) | Up to 3 Years

SECONDARY OUTCOMES:
Overall Response Rate (ORR) as assessed by the investigator | Up to 3 Years

CONTACTS AND LOCATIONS:
Overall Officials: Jason Wu, Study Chair — Suzhou Zelgen Biopharmaceuticals Co.,Ltd
Locations (1):
- Zhejiang Cancer Hospital, Zhejiang, Hangzhou, China